CLINICAL TRIAL: NCT06253520
Title: A Phase Ib Clinical Trial to Evaluate the Administration of Autologous T-cells Genetically Engineered to Express Receptors Reactive Against KRAS Mutations in Conjunction With a Vaccine Directed Against These Antigens in Participants With Metastatic Cancer
Brief Title: Autologous T-cells Genetically Engineered to Express Receptors Reactive Against KRAS Mutations in Conjunction With a Vaccine Directed Against These Antigens in Participants With Metastatic Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10001662; 001662-C
Record Dates: First submitted 2024-02-09; First posted 2024-02-12 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10-16

CONDITIONS: Metastatic Solid Cancers; Colorectal Cancer; Breast Cancer; Non-Small Cell Lung Cancer; Gastrointestinal Cancer; Ovarian Cancer; Genitourinary Cancer
Keywords: KRAS Mutations; Gene Therapy; Cell Therapy; Immunotherapy; Vaccine
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Gastrointestinal Neoplasms; Ovarian Neoplasms; Urogenital Neoplasms | interventions — aldesleukin; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/ KRAS TCR + vaccine (Experimental): Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine + KRAS TCR-Transduced PBL + high-dose aldesleukin + vaccine (Day 0, weeks 4 and 8 and at week 12 (if no progression)
  Interventions: Drug: Aldesleukin; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: KRAS TCR-Transduced PBL; Biological: GRT-C903/GRT-R904

INTERVENTIONS:
Drug: Aldesleukin — Aldesleukin 600,000 IU/kg IV (based on total body weight) over 15 minutes approximately every 8 hours beginning within 24 hours of cell infusion and continuing for up to 4 days (maximum 10 doses). Patients in Cohort 3 may receive 72,000 IU/kg IV.
Drug: Fludarabine — Days -7 to -3: Fludarabine 25 mg/m2/day IVPB daily over 30 minutes for 5 days.
Drug: Cyclophosphamide — Days -7 and -6: Cyclophosphamide 60 mg/kg/day x 2 days IV in 250 mL D5W infused simultaneously with mesna 15 mg/kg/day over 1 hour x 2 days.
Biological: KRAS TCR-Transduced PBL — Day 0: Cells will be infused intravenously (IV) over 20-30 minutes (2-4 days after the last dose of fludarabine).
Biological: GRT-C903/GRT-R904 — Day 0 (GRT-C903): Injection of 1.0 mL at each of 2 bilateral vaccine injections. Weeks 4, 8 and 12 (as applicable, GRT-R904): Injection of 0.25 mL of diluted GRT-R904 at each of 2 bilateral vaccine injections

SUMMARY:
Background:

Many cancer cells produce substances called antigens that are unique to each cancer. These antigens stimulate the body s immune responses. One approach to treating these cancers is to take disease-fighting white blood cells from a person, change those cells so they will target the specific proteins (called antigens) from the cancer cells, and return them to that person s blood. The use of the white blood cells in this manner is one form of gene therapy. A vaccine may help these modified white cells work better.

Objective:

To test a cancer treatment that uses a person s own modified white blood cells along with a vaccine that targets a specific protein.

Eligibility:

Adults aged 18 to 72 years with certain solid tumors that have spread after treatment.

Design:

Participants will undergo leukapheresis: Blood is removed from the body through a tube attached to a needle inserted into a vein. The blood passes through a machine that separates out the white blood cells. The remaining blood is returned to the body through a second needle.

Participants will stay in the hospital for 3 or 4 weeks. They will take chemotherapy drugs for 1 week to prepare for the treatment. Then their modified white cells will be infused through a needle in the arm. They will take other drugs to prevent infections after the infusion.

The vaccine is injected into a muscle; participants will receive their first dose of the vaccine on the same day as their cell infusion.

Participants will have follow-up visits 4, 8, and 12 weeks after the cell infusions. They will receive 2 or 3 additional doses of the boost vaccine during these visits.

Follow-up will continue for 5 years, but participants will need to stay in touch with the gene therapy team for 15 years.

...

DETAILED DESCRIPTION:
Background:

* The majority of cancer deposits from patients with melanoma or solid epithelial cancers contain tumor infiltrating lymphocytes (TIL) that can recognize unique mutated neoantigens expressed by the cancer.
* Administration of autologous TIL to patients with metastatic melanoma can mediate complete durable regression in up to 24% of patients with metastatic melanoma. The administration of TIL from patients with solid epithelial cancers mediate far fewer clinical responses probably because the frequency of these anti-tumor T cells in solid epithelial cancers is very low (often less than 0.1%).
* We have developed approaches to adoptive cell transfer (ACT) therapy that involves isolating T-cell receptors (TCR) that recognize mutated cancer neoantigen. These TCRs are transduced into autologous peripheral lymphocytes to express these TCRs with high efficiency. These neoantigen TCR gene-modified cells can recognize and destroy the autologous cancer in vitro.
* In a single patient with chemo-refractory metastatic colon cancer, we identified a rare population of neoantigen reactive TIL targeting the KRAS G12D hotspot mutation and administration of these TIL mediated a near-complete regression of all metastatic disease now lasting over 5 years. The administration of cells genetically modified to express anti KRAS G12D receptors obtained from this patient have now been used to mediate regression of metastatic pancreatic cancer in a patient containing a G12D mutation. Using targeted screening and in vitro sensitization of PBL and TIL, we have now identified a library of TCRs capable of recognizing the KRAS G12D or KRAS G12V shared mutations restricted by a variety of Class I or Class II MHC restriction elements.
* In murine experiments utilizing T-cell receptors against mutated antigens, we have shown that cells bearing these receptors are far more effective in mediating anti-tumor responses against established tumors when cell administration is combined with a vaccine targeting the same antigen targeted by the T cells.
* Gritstone bio has developed a prime boost adenoviral/mRNA vaccine targeting KRAS G12D and G12V shared mutations.
* The clinical protocol described here will treat participants with chemorefractory solid cancers that express G12D or G12V KRAS mutations using the adoptive transfer of autologous lymphocytes transduced with genes encoding TCRs that recognize these mutations in conjunction with the administration of an anti-KRAS vaccine.

Objectives:

-Primary objective:

--Determine the safety and efficacy of administering autologous T cells transduced to express receptors targeting KRAS G12D or G12V mutations in conjunction with an anti-KRAS vaccine to participants with metastatic solid cancers that contain KRAS G12D or G12V mutations.

Eligibility:

-Participants must be/have:

* Age >= 18 years and <= 72 years
* Metastatic cancer that expresses either the KRAS G12D or KRAS G12V hotspot mutation for which the Surgery Branch has identified TCRs capable of recognizing these antigens with appropriate MHC restriction.
* Evaluable solid cancer that has recurred following standard systemic therapy.
* Adequate basic laboratory values.
* No concurrent major medical illnesses or any form of immunodeficiency.

Design:

* Participants who have cancers demonstrated to contain KRAS G12D or G12V genetic mutations in the autologous cancer will be included.
* T-cell receptors that recognize KRAS G12D or G12V mutations will be inserted into participant PBL and used for cell transfer immunotherapy. Participants will also receive a KRAS prime-boost vaccine that expresses G12D and G12V hotspot mutation epitopes.
* Participants will be enrolled into one of four cohorts: (1) G12D KRAS mutations treated with TCRs recognizing these mutations restricted by Class I MHC molecules, (2) G12D KRAS mutations treated with TCRs recognizing these mutations restricted by Class II MHC molecules, (3) G12V KRAS mutations treated with TCRs recognizing these mutations restricted by Class I MHC molecules, (4) G12V KRAS mutations treated with TCRs recognizing these mutations restricted by Class II MHC molecules.
* Clinical and immunologic responses will be evaluated about 4-6 weeks after cell infusion and periodically thereafter.
* It is anticipated that approximately 3 participants may enroll on the trial each month. There will be an initial limit of 21 evaluable participants per cohort for a total of 84 evaluable participants. Thus, the initial accrual may be completed in approximately 3 years. Any group moving to a second-stage evaluation would accrue an additional 29 evaluable participants over approximately two years for a potential total of 200 evaluable participants.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants with an appropriate HLA match for available Surgery Branch KRAS TCRs with evaluable metastatic solid cancer (e.g., gastrointestinal, genitourinary, breast, ovarian, non-small cell lung cancer (NSCLC) and other solid cancers) with known KRAS G12V or G12D mutation.
* Confirmation of diagnosis of cancer by the NCI Laboratory of Pathology.
* Refractory to standard systemic therapy. Specifically:

  * Participants with metastatic colorectal cancer must have received oxaliplatin and/or irinotecan.
  * Participants with breast and ovarian cancer must have received at least two systemic treatments.
  * Participants with NSCLC must have received at least one platinum-based chemotherapy regimen and at least one FDA-approved targeted treatment (when appropriate).
  * Participants with other solid tumors must have received at least one prior line of systemic treatment or have declined standard treatment.
  * Participants with three (3) or fewer brain metastases that are < 1 cm in diameter each and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for one month after treatment for the participant to be eligible. Participants with surgically resected brain metastases are eligible.
* Age >= 18 years and <= 72 years.
* Clinical performance status of ECOG 0 or 1.
* Individuals of child-bearing potential (IOCBP) must agree to use highly effective contraception (hormonal, intrauterine device [IUD, abstinence, surgical sterilization starting at the time of study entry, for the duration of study therapy, and 12 months after the last dose of combined chemotherapy

Participants who can father a child must agree to use an effective method of contraception (barrier, surgical sterilization, abstinence) for the duration of the study treatment and for 4 months after the last dose of combined chemotherapy. We also will recommend participants that can father children with partners of childbearing potential to ask their partners to be on highly effective birth control (hormonal, intrauterine device (IUD), surgical sterilization).

NOTE: IOCBP is defined as any person who has experienced menarche and who has not undergone successful surgical sterilization or who is not postmenopausal.

NOTE: Certain malignancies may secrete hormones that produce false positive pregnancy tests. Serial blood testing (e.g. HCG measurements) and/ or ultrasound may be performed for clarification.

* Participants must have serology results as follows:

  * Seronegative for HIV antibody.
  * Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then participant must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
* Adequate organ and marrow function as defined below:

  --Hematology:
  * ANC > 1000/mm^3 without growth factor support
  * WBC >= 2500/mm^3
  * Platelet count (Bullet) 80,000/mm3
  * Hemoglobin > 8.0 g/dL. Subjects may be transfused to reach this cut-off.
* Chemistry:
* Serum ALT/AST <= 5.0 x ULN
* Serum creatinine <= 1.6 mg/dL
* Total bilirubin <= 2.0 mg/dL, except in participants with Gilbert s Syndrome, who must have a total bilirubin < 3.0 mg/dL.
* Participants must have completed any prior systemic therapy at the time of enrollment.

NOTE: Participants may have undergone minor surgical procedures or limited field radiotherapy within the four weeks prior to enrollment, as long as related major organ toxicities have recovered to grade 1 or less.

* For participants with NSCLC or lung metastases, more than two weeks must have elapsed since any prior palliation for major bronchial occlusion or bleeding at the time the patient receives the preparative regimen, and patient s toxicities must have recovered to a grade 1 or less.
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Willing to sign a durable power of attorney.
* Participants must be co-enrolled on protocol 03-C-0277.

EXCLUSION CRITERIA:

* Participants who are pregnant or nursing because of the potentially dangerous effects of the treatment on the fetus or infant.
* Any form of secondary immunosuppression.
* Active systemic infections requiring anti-infective treatment, coagulation disorders, or any other active or uncompensated major medical illnesses.
* For participants with NSCLC or lung metastases, any major bronchial occlusion or bleeding not amenable to palliation.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease and AIDS).
* History of major organ autoimmune disease.
* Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Participants who have decreased immune-competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
* History of severe immediate hypersensitivity reaction to cyclophosphamide, fludarabine, aldesleukin or vaccines.
* Clinically significant participant history which in the judgment of the Principal Investigator (PI) would compromise the participants ability to tolerate high-dose aldesleukin.
* History of coronary revascularization or ischemic symptoms.
* For select participants with a clinical history prompting cardiac evaluation: last known LVEF <= 45%.
* For select participants with a clinical history prompting pulmonary evaluation: known FEV1 <= 50% predicted.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2031-06-15 (Estimated); Study Completion 2033-06-15 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) and/ or partial response (PR) | Response assessed at 4, 8, 12 and 20 weeks post-cell infusion, every 3 months x3, every 6 months x 2 years
  Clinical response rate ([PR+CR]/evaluable participants) will be determined and reported along with the corresponding 95% two-sided confidence interval.
Safety | All adverse Events (AE) per CTCAE v5.0, by type and grade of toxicity, from first dose through 4 weeks after the last treatment
  Safety and tolerability will be analyzed by reporting the number of patients experiencing toxicity, classified by type and grade to the experimental regimen. Adverse events assessed per CTCAE version 5.

SECONDARY OUTCOMES:
Safety | From study treatment initiation up to 4 weeks after the last study treatment
  The number of participants with toxicity of grade 3 or higher related to the KRAS-TCR transduced cells or vaccine, according to type of toxicity. Adverse events assessed per CTCAE version 5.

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared. All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review and/or will involve genomic data sharing.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001662-C.html